CLINICAL TRIAL: NCT05676606
Title: Official Title: Remote 1-minute Single-lead Electrocardiogram (ECG) Monitoring for Cardiotoxicity Detection in Patients With the First Diagnosed Cancer After the First Cycle of Polychemotherapy
Brief Title: Cardiotoxicity Monitoring With Single-lead Electrocardiogram
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FZ 01
Record Dates: First submitted 2022-12-22; First posted 2023-01-09 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2023-01

CONDITIONS: Cardiotoxicity
Keywords: 1-minute; single-lead ECG; cardiotoxicity; chemotherapy
MeSH Terms: conditions — Cardiotoxicity | interventions — Electrocardiography

STUDY DESIGN:
Intervention Model Description: a group of chemotherapy-naive patients with first time diagnosed various kinds of tumors, planned for the first cycle polychemotherapy treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- monitoring group (Experimental): a group of chemotherapy-naive patients with first time diagnosed various kinds of tumors, planned for the first cycle polychemotherapy treatment.
  Interventions: Device: Remote 1-minute single-lead electrocardiogram (ECG) monitoring in cancer patients after the first polychemotherapy cycle.

INTERVENTIONS:
Device: Remote 1-minute single-lead electrocardiogram (ECG) monitoring in cancer patients after the first polychemotherapy cycle. — Recording of the ECG using smart-phone at rest, 15 minutes before registering ECG patient should not smoke,having tea, coffee, alcohol. During the ECG recording hands should be fixed to avoid poor quality. Patient sitting on a char with tow hands fixed on a table holding electrocardiograph with index fingers placed at the ECG electrode (left) and at the photoplethysmograph sensor(right).ECG signals are recorded from the fingers using first standard ECG lead. After registration, all ECG and photoplethysmography data will be sent to the server. The data will be automatically compared with a standard for data quality, after that the data will be sent to cardiologist. If quality will be not sufficient, the data will be deleted and the doctor will contact the patient to solve the quality issue. Thereafter, the parameters will be carried out by cardiologist, on the basis of which value of ECG monitoring will be estimated.

SUMMARY:
This research is a multi-center prospective cohort interventional study aimed to determinate the capabilities of remote 1-minute single-lead electrocardiogram monitoring for cardiotoxicity detection, during two- three weeks (depending on the scheme of polychemotherapy) after the first cycle of polychemotherapy in patients with the first diagnosed cancer.

DETAILED DESCRIPTION:
The study planned to include 130 patients and will be conducted in three stages:

Stage one - screening (the day before chemotherapy treatment):

1. Signing a voluntary informed consent to participate in the study;
2. Clinical examination; Questioning: finding out the complaints. Anamnesis morbid: investigation of the history of cardiovascular diseases (the presence of hypertension, ischemic heart disease, diabetes mellitus, congenital heart disease, heart surgery in the past).

   Anamnesis vitae: investigation of the history of patient's life (place of birth, development in childhood and adolescence, tobacco smoking, consumption of alcohol beverage, narcotic drugs, sleeping pills and sedatives, strong tea and coffee).
3. Assessment patient's risk profile according to the cardiotoxicity risk assessment scale for treatment of tumors (C.M. Larsen assessment scale 2014).

   Risk level-the sum of points of all risks ((1) the risk associated with the specific chemotherapy that will be received and (2) the risk related to co-existing cardiac risk factors, age and sex of patients), these factors can be used to generate a risk score: >6 points-very high risk, 5-6 points - high risk; 3-4 points- intermediate risk; 1-2 points-rare risk;
4. All patients included in the study will be registered in single-lead ECG server base and will be trained to use single-lead electrocardiograph themselves. Before starting chemotherapy, each patient will record an 1-minute single-lead ECG.
5. Instrumental examination: transthoracic echocardiography with assessment of left ventricular ejection fraction (LVEF) and speckle-tracking global longitudinal strain (GLS), standard 12-lead electrocardiography;
6. Laboratory testing: cardiac serum biomarkers-n-terminal pro b-type natriuretic peptide(NT-proBNP), highly sensitive troponin I.

Stage two - interim home control (during 2-3 weeks after first cycle of the chemotherapy):

During this period, patients will registrate a single-lead electrocardiogram by themselves using single-lead ECG device, every day the patient should do at least 5 ECG records. The data will be sent to the server database, where cardiologist will check it for pathology, poor quality and will contact patients, if needed.

Stage three - final control (after first course of the chemotherapy):

1. Patients' clinical examination, complaints registration;
2. Instrumental examination: transthoracic echocardiography with assessment of left ventricular ejection fraction (LVEF) and speckle-tracking global longitudinal strain (GLS), standard 12-lead electrocardiography;
3. Laboratory testing:cardiac serum biomarkers -n-terminal pro b-type natriuretic peptide (NT-proBNP), highly sensitive troponin I);
4. Evaluation of outcomes,depending on the patient's complaints, the results of instrumental and biochemical test methods carried out. The patient will be given recommendations necessary for their cardiovascular disorders correction;
5. Database compilation and statistical processing.

ELIGIBILITY:
1. Inclusion Criteria:

   * chemotherapy-naive patients with first time diagnosed various kinds of tumors, planned for the first cycle polychemotherapy treatment over 18 years old
   * Written informed consent to participate in the study.
   * Patients without decompensation of cardiovascular diseases
2. Non-inclusion criteria:

   * Pregnancy;
   * Severe hepatic and\or renal failure(glomerular filtration rate below 30 (ml\min\1.732) Cockcroft-Gault, Child-Pugh score less than 6 points;
   * Radiation therapy and\or any surgical treatment in last 30 days.
   * Heart failure with left ventricular ejection fraction< 50 %, III-IV functional class New York Heart Association Functional Classification (NYHA)
   * Cardiac arrhythmias - permanent form of atrial fibrillation\flutter, atrioventricular block (AV block) II-III degree
   * Congenital or acquired heart valve disease
   * Patients with impaired motor function or tremor of the upper limb. As well as patients with severe cognitive impairments
   * Patients with a minimum life expectancy of less than 1 month
3. Exclusion Criteria:

   * Refusal to further participate in the study;
   * Non-compliance to the therapy regimen.
   * Poor quality ECG, poor echocardiography visualization,detection a defect of the preanalytical stage of the blood biochemical analysis (hemolysis, non-compliance with the temperature regime, long-term transportation, long-term storage, long-term or repeated centrifugation).
   * Development of other toxicity during chemotherapy treatment, which might prevents the evaluation of the study results

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-05-25 (Actual)

PRIMARY OUTCOMES:
Severe asymptomatic cancer-therapy related cardiac dysfunction | Up to one month after the first cycle of chemotherapy treatment
  Left ventricular ejection fraction reduction (LVEF) to < 40% .
Moderate asymptomatic cancer-therapy related cardiac dysfunction | Up to one month after the first cycle of chemotherapy treatment
  LVEF reduction by ≥10 percentage points to an LVEF of 40-49% or new LVEF reduction by < 10 percentage points to an LVEF of 40-49% and either new relative decline in GLS by >15% from baseline or new rise in cardiac biomarkers;
Mild asymptomatic cancer-therapy related cardiac dysfunction | Up to one month after the first cycle of chemotherapy treatment
  LVEF ≥ 50% and new relative decline in GLS by >15% from baseline and/or new rise in cardiac biomarkers.
Chemotherapy-induced atrial fibrillation\ flutter. | Up to one month after the first cycle of chemotherapy treatment
  Rhythm with no discernible repeating P waves and irregular RR intervals is diagnosed on an standard 12-lead ECG or a single-lead ECG tracing of ≥ 30 s recording
Chemotherapy- induced atrioventricular block I-III degrees | Up to one month after the first cycle of chemotherapy treatment
  * First-degree atrioventricular block, on ECG, this is defined by a PR interval greater than 200 mc
  * Second-degree atrioventricular block; not all P-waves are followed byQRS complexes.
  Second-degree atrioventricular blockMobitz type I- this manifest on the ECG as gradual increase of PR interval before a block of QRS complexes occurs.
  Second-degree atrioventricular blockMobitz type II-the block of QRS complexes occurs without gradual increase of PR interval.
  • Third degree atrioventricular block- on the ECG P-waves have no relation to the QRS complexes.
Chemotherapy-induced QTc interval prolongation: | Up to one month after the first cycle of chemotherapy treatment
  QTc> 500 ms and\or QTc> 60 ms deviation from baseline.
Chemotherapy-induced arterial hypertension: | Up to one month after the first cycle of chemotherapy treatment
  Steady increase in systolic arterial blood pressure ≥140 mmHg and/or diastolic ≥90 mmHg in period after chemotherapy.
Chemotherapy-induced arterial hypotension. | Up to one month after the first cycle of chemotherapy treatment.
  Steady decrease in systolic arterial blood pressure ≤ 100 mmHg and/or diastolic ≤ 90 mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Kopylov, MD, Study Director — I.M. Sechenov First Moscow State Medical University (Sechenov University)
Locations (1):
- I.M. Sechenov First Moscow State Medical University (Sechenov University), Moscow, Russia

IPD SHARING:
Plan to Share IPD: No
local ethics committee prohibits disclosure patients' information Information can be provided upon official request addressed to the principal investigator